CLINICAL TRIAL: NCT03925805
Title: Quality of Life in Patients With Chronic Disease
Acronym: QAPICHE
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Principal Investigator, VakgroepVolksgezondheidEnEerstelijnszorg, Public Health and Primary Care, University Ghent
Other Study IDs: B670201939629
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Chronic Disease; Quality of Life; Cardiovascular Diseases; Diabetes; Mental Disorder; Musculoskeletal Disease
MeSH Terms: conditions — Chronic Disease; Cardiovascular Diseases; Diabetes Mellitus; Mental Disorders; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic disease: Cardiovascular disease (including diabetes), mental disease, musculoskeletal disease

SUMMARY:
To improve HRQoL in patients with chronic diseases, a comprehensive understanding of the association between HRQoL and chronic diseases is vital. Therefore, the aim of the study is to provide a profound insight in HRQoL outcomes and its determinants in chronically ill patients, with a focus on multimorbidity and socio-economic status in a primary care setting.

DETAILED DESCRIPTION:
A primary care based cross-sectional study will be conducted to investigate HRQoL in adult patients with chronic diseases in Flanders (Belgium).

To achieve the research aims, multiple linear regression models will be conducted assessing several key predictors associated to HRQoL as primary outcome. The regression models should allow for controlling the effect of main confounders (e.g., sex, age, educational attainment), and for including interaction terms with psychosocial variables. A sample size calculation showed that the minimum required sample for a multiple regression study including 10 predictors with a medium anticipated effect size was 118, given a desired statistical power level of 80% and a probability level of 5%. The sample size was increased with 50% to allow for testing interaction effects. This study has three clusters of disease groups (cardiovascular disorders, mental disorders, and musculoskeletal disorders), therefore stratified analyses require a triple sample size. Hence, an a priori sample size of minimum 531 participants is targeted. This sample size will also widely cover analyzing clinically relevant differences between a number of chronic disease subgroups. Based on the conclusions of a systematic review by Norman et al. (2003), the clinically relevant difference will be set at a half standard deviation which appears to be the threshold of discrimination for changes in HRQoL for NCDs. Using a statistical power level of 80% and a probability level of 5%, information on 76 patients per disease cluster is needed 1) to assess the HRQoL (based on SF-36) in each patients group with a 5% precision and 2) to allow for comparisons across groups.

Patient recruitment will be organized through general practitioners (GP) and community health centers across Flanders (Belgium). First, a number of GP practices located across urban and rural regions willing to participate in this study will be identified through a convenience sample based on their contact with a LOK group (Local Quality Group). This is a group of colleagues, doctors or pharmacists-biologists, who share and critically assess their medical practices (peer review) in order to improve the quality of care. GPs willingness to cooperate in the study will be asked at the LOK group meeting. In this meeting, the researchers will briefly present the study. Afterwards, interested GPs will be visited by the researchers at their practice with more detailed information about the study and they will receive the paper questionnaires. GPs will be asked to identify patients within their practice after validation of the eligibility criteria. GPs will explain briefly the purposes of the study to the patients and invite them to participate through voluntary response sample.

A paper-based questionnaire, including informed consent, will be distributed to the participant by the GP at consultation. The questionnaire will be filled in by the patient at home. Afterwards, the patient can return the questionnaire to the researchers for free via a prepaid envelope or the questionnaire can be given back to the GP at later consultation. The questionnaire will take 30 minutes to gather patient information and research outcomes. The GPs will receive in advance detailed information by the researcher to ensure the aim of the study and the data collection process are understood. Due to practical restrictions, home visits for fulfilling the questionnaires was not achievable in this study.

Descriptive statistics will be reported in order to describe the sample of the study participants. Means, standard deviations, median, and percentages for the continuous variables and frequency tables for categorical variables will be displayed. Socio-demographic differences between study participants will be tested with the appropriate test.

Exploratory data analysis will be performed both for the continuous variables as well as the categorical variables. T-tests and one-way analysis of variance will be reported to compare groups when normal distribution is applicable. Non-parametric tests will be used when variables are not normally distributed. A p-value of 0.05 will be considered as statistically significant. Furthermore, multiple linear regression models will be conducted assessing several main determinants, such as multimorbidity and SES, associated to HRQoL as main outcome parameter. Furthermore, the study results will be validated against the HRQoL data collected in the Health Interview Survey with the aim to predict future HRQoL burden.

ELIGIBILITY:
Inclusion Criteria:

* Study participants have to be adults (aged 18 years or older).
* Study participants need to be medically diagnosed with one (or more) diseases of the following three non-infectious disease groups, in various degrees of severity:cardiovascular disorders (including diabetes), mental disorders, and musculoskeletal disorders.
* Study participants must have been followed by their general practitioner for at least six months.
* Study participants must have good understanding of Dutch to be able to complete the questionnaire and to give informed consent.

Exclusion Criteria:

* Study participants with a major cognitive impairment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any chronic disease that fits in the three major disease groups, can be included. The selection of these specific disease groups was determined by a literature search. It was found that these disease groups result in a lower quality of life compared to other diseases.
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (EQ-5D-5L) | Measured at one time point (inclusion)
  Health-related quality of life will be measured using the EuroQol Five Dimensions (EQ-5D). The EQ-5D-5L is a valid extension of the 3-level questionnaire. It can be defined as a standardized non-disease specific value-based instrument to describe and value health-related quality of life. The instrument consists of two components: the EQ-5D descriptive system and the EQ visual analogue scale (EQ-VAS).The first part consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response categories (no problems, slight problems, moderate problems, severe problems, and extreme problems), from which a single EQ-5D index score can be calculated ranging from 0 (dead) to 1 (perfect health). The EQ-VAS measures one's self-perceived health today on a vertical scale from 0 (worst imaginable health) to 100 (best imaginable health) on which participants have to indicate their current health.
Self-perceived health status (SF-12) | Measured at one time point (inclusion)
  This study will use the 12-item Short Form Health Survey (SF-12) as a generic subjective or self-perceived health status instrument to assess patient's functional health and well-being whereas both physical and mental functioning components can be measured. This study makes use of the 12-item version instead of the 36-item version, because it can be completed in a shorter time. This instrument contains 12 items including eight domains (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health) which can be easily completed in five minutes. The summary scores, on a scale from 0 to 100, will be calculated to represent physical (Physical Component Summary score) and mental functioning (Mental Component Summary score). Higher scores indicate better self-perceived health status. The SF-12 has been confirmed as a valid and reliable instrument for measuring health perception in a general population for primary care.

SECONDARY OUTCOMES:
Sense of coherence (SOC-13) | Measured at one time point (inclusion)
  Sense of coherence will be measured using the brief Antonovsky's Sense of Coherence Scale (SOC) which contains 13 items covering three dimensions: comprehensibility (the extent to which events are perceived as making sense, that they are ordered, consistent and structured), manageability (the extent to which a person feels he/she can cope), and meaningfulness (how much one feels that life makes sense and challenges are worthy of commitment). Responses are reported by a semantic scale ranging from one (never or very seldom) to seven points (very often). SOC scores range from 13 to 91, and a higher score indicates higher SOC.
Self-efficacy (GSES) | Measured at one time point (inclusion)
  General self-efficacy will be measured using the General Self-Efficacy Scale (GSES). The GSES is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. The total score is calculated by the sum of all items. Scores range between 10 and 40, with higher scores indicating more self-efficacy.
Health literacy (HLS-EU-Q6) | Measured at one time point (inclusion)
  The HLS-EU-Q6 will be used as a short scale of the European Health Literacy Survey (HLS-EU-Q). This tool consists of 6 items addressing self-reported difficulties in accessing, understanding, appraising and applying information in tasks concerning decision-making in health care, disease prevention, and health promotion. Responses are reported from one (very difficult) to four (very easy). The scale score varies between 1 and 4, with higher scores indicating better health literacy.
Patient enablement (PEI) | Measured at one time point (inclusion)
  The Patient Enablement Instrument (PEI) focuses on the impact of a clinical consultation for an acute or chronic disease in primary care on a patient's self-perceived ability to understand and cope with health issues and disease. It consists of six questions that reflect patient enablement. The responses are scored on a three-point scale (same or less/not applicable = 0, better/more = 1, and much better/much more = 2). The total PEI score ranges between 0 and 12 to indicate low (0-4), medium (score 5-9), and high enablement (10-12).
Social support (F-SozU) | Measured at one time point (inclusion)
  Social support will be measured using the 6-item shortened version of the Social Support Questionnaire (F-SozU). This valid and reliable instrument is well accepted in epidemiologic contexts to assess social support in the general population. Responses are rated on a five-point Likert scale, ranging from 1 (does not apply) to 5 (exactly applicable). The total range is from 0 to 30 with higher values representing higher perceived and received social support.
Multimorbidity | Measured at one time point (inclusion)
  Multimorbidity will be measured by a self-developed list based on the MultiMorbidity Questionnaire (MM-21), and documents 24 self-reported chronic conditions in primary care. Participants have to indicate for each condition 'yes' or 'no', 'yes' may only be filled in for the conditions that have been confirmed by a doctor or for which the participant is taking prescribed drugs.
Symptoms (HADS) | Measured at one time point (inclusion)
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item brief self-reported instrument to determine possible presence of anxiety and depressive states. The HADS compromises two scales, each consisting of seven items. A maximum score of 21 can be achieved per scale. The higher the overall score, the higher levels of anxiety and depression.
Illness perception (IPQ-B) | Measured at one time point (inclusion)
  The brief Illness Perception Questionnaire (IPQ-B) will be used for assessing patients' cognitive and emotional representations of their illness including consequences, timeline, personal control, treatment control, identity, coherence, concern, emotional response, and causes. The questionnaire uses a scale from 0 to 10 to assess cognitive illness representations (IPQcognitive, item 1-5), emotional representations (IPQemotional, item 6 and 8), and illness comprehensibility (IPQcomprehensibility, item 7). A low score on items number 1,2,5,6 and 8 indicates that the illness is perceived as benign while a low score on the items 3, 4 and 7 indicates that the illness is perceived as threatening. By reversing these three items it is possible to compute an overall score. A higher score reflects a more threatening view of the illness.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine De Smedt, PhD, Principal Investigator — University Ghent
Locations (1):
- Lisa Van Wilder, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided